CLINICAL TRIAL: NCT01367665
Title: A Single Arm, Open-label, Phase II, Multicentre Study, to Assess the Safety of Vismodegib (GDC-0449) in Patient With Locally Advanced or Metastatic Basal Cell Carcinoma (BCC)
Brief Title: STEVIE: A Study of Vismodegib in Patients With Locally Advanced or Metastatic Basal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO25616; 2011-000195-34 (EudraCT Number)
Record Dates: First submitted 2011-05-30; First posted 2011-06-07 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-03

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

ARMS (2):
- Vismodegib - Locally Advanced (Experimental): Participants received vismodegib 150 mg orally once a day until one of the following occurs: Disease progression, intolerable toxicity most probably attributable to vismodegib, consent withdrawal, death, study termination by the Sponsor, or other reason deemed by the Investigator. vismodegib: 150 mg once daily until disease progression or unacceptable toxicity
  Interventions: Drug: vismodegib
- Vismodegib - Metastatic (Experimental): Participants received vismodegib 150 mg orally once a day until one of the following occurs: Disease progression, intolerable toxicity most probably attributable to vismodegib, consent withdrawal, death, study termination by the Sponsor, or other reason deemed by the Investigator. vismodegib: 150 mg once daily until disease progression or unacceptable toxicity
  Interventions: Drug: vismodegib

INTERVENTIONS:
Drug: vismodegib — 150 mg once daily until disease progression or unacceptable toxicity

SUMMARY:
This single-arm, open-label, multi-center study will evaluate the safety and efficacy of vismodegib (GDC-0449) in patients with locally advanced or metastatic basal cell carcinoma. Patients will receive oral doses of vismodegib 150 mg once daily until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Metastatic or locally advanced basal cell carcinoma considered inoperable or that surgery is contraindicated and radiotherapy is contraindicated or inappropriate
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2

Exclusion Criteria:

* Concurrent anti-tumor therapy
* Completion of the most recent anti-tumor therapy less than 21 days prior to the initiation of treatment
* Uncontrolled medical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1232 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (181):
- Inst. de Oncologia Angel H. Roffo ; Servicio de Oncologia, Buenos Aires, Argentina
- Australia (4):
  - Premier Specialists, Kogarah, New South Wales
  - Skin and Cancer Foundation Australia, Westmead, New South Wales
  - CMAX A division of IDT Australia Limited, Adelaide, South Australia
  - Skin & Cancer Foundation, Carlton, Victoria
- Austria (4):
  - LKH Graz; Abteilung für allgemeine Dermatologie, Graz
  - LKH Salzburg; Universitätsklinik für Dermatologie, Salzburg
  - Landesklinikum St. Pölten, Sankt Pölten
  - Medizinische Universität Wien; Univ.Klinik für Dermatologie, Vienna
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Bosnia and Herzegovina (2):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - Clinic of Oncology, University Clinical Center Sarajevo, Sarajevo
- Brazil (3):
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Bulgaria (2):
  - District Oncology Dispensary; Department for Oncology and Dermatology, Plovdiv
  - National Specialized Hospital for Active Oncology Treatment; Dermatology Clinic, Sofia
- Canada (6):
  - Western Canada Dermatology Institute, Edmonton, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - London Regional Cancer Centre, London, Ontario
  - Dr. Nowell Solish Cosmetic Dermatology, Toronto, Ontario
  - Victoria Park MediSpa, Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec Metropolitain (CRDQ), Québec
- Colombia (5):
  - Inst. Nacional de Cancerologia; Clinica de Seno, Bogotá
  - Riesgo De Fractura; Rheumatology, Bogotá
  - Hemato Oncologos S.A., Cali
  - Hospital Pablo Tobon Uribe, Medellin-Antioquia
  - Reumalab Sas; Rheumatology, Medellín
- Clinical Hospital Sisters of Mercy, Zagreb, Croatia
- Czechia (7):
  - Nemocnice Ceske Budejovice, České Budějovice
  - Fakultni Nemocnice Hradec Kralove; Dept of Radiotherapy & Oncology, Hradec Králové
  - Fakultní nemocnice Ostrava; Kožní oddělení, Ostrava
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni Thomayerova Nemocnice; Onkologicke Oddeleni, Prague
  - Fakultni nemocnice v Motole, Prague
- Herlev Hospital; Onkologisk afdeling, Herlev, Denmark
- Finland (2):
  - Helsinki University Central Hospital; Skin & Allergy Hospital, Helsinki
  - Kuopion yliopistollinen sairaala, Kuopio
- France (11):
  - Hopital Saint Andre CHU De Bordeaux; Dermatologie, Bordeaux
  - Hopital Ambroise Pare; Sce Dermatologie, Boulogne-Billancourt
  - Chu Site Du Bocage;Dermatologie, Dijon
  - Hopital Claude Huriez; Sce Dermatologie, Lille
  - Hopital Timone Adultes; Dermatologie, Marseille
  - Hopital Saint Eloi; CHU de Montpellier; Svc de Dermatologie, Montpellier
  - Hopital Hotel Dieu Et Hme; Clinique Dermatologique, Nantes
  - Hopital Saint Louis; Dermatologie 1, Paris
  - Centre Hospitalier Lyon Sud; Dermatologie, Pierre-Bénite
  - Hôpital Larrey Université Paul Sabatier; Service Dermatologie, Toulouse
  - Institut Gustave Roussy; Comite 5, Villejuif
- Germany (31):
  - Charité Campus Mitte; Hauttumorcentrum Charité (HTCC); Klinik für Dermatologie, Venerologie und Alle, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Elbekliniken Buxtehude; Klinik für Dermatologie, Buxtehude
  - Klinik der Uni zu Köln; Klinik & Poliklinik fuer Dermatologie & Venerologie, Cologne
  - Klinikum Dortmund gGmbH Klinikzentrum Mitte, Dortmund
  - Universitätsklinikum "Carl Gustav Carus"; Klinik und Poliklinik für Dermatologie, Dresden
  - Universitätsklinikum Düsseldorf; Hautklinik, Düsseldorf
  - HELIOS Klinikum Erfurt; Klinik für Dermatologie & Allergologie, Erfurt
  - Universitätsklinikum Essen, Essen
  - Klinik Johann Wolfgang von Goethe Uni; Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt
  - Universitätsklinikum Freiburg Universitäts-Hautklinik, Freiburg im Breisgau
  - Universitätsmedizin Greifswald; Klinik für MKG-Chirurgie und Plastische Operationen, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf Zentrum f.Innere Medizin Klinik f.Dermatologie, Hamburg
  - Medizinische Hochschule Hannover; Klinik für Dermatologie, Allergologie und Venerologie, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum am Gesundbrunnen; Tumorzentrum, Heilbronn
  - Klinikum Kassel; Hautklinik, Kassel
  - UNI-Klinikum Campus Kiel Klinik f.Dermatologie Tagesklinik f.Dermatologie, Kiel
  - Klinikum d.Stadt Ludwigshafen Hautklinik, Ludwigshafen
  - Uni Schleswig-Holstein; Klinik für Dermatologie, Allergologie und Venerologie (Hautklinik), Lübeck
  - Universitätsklinikum Magdeburg; Hautklinik; Klinik für Dermatologie und Venerologie, Magdeburg
  - Klinikum Mannheim Klinik fuer Dermatologie, Venerologie und Allergologie, Mannheim
  - Universitätsklinikum Marburg Klinik f. Dermatologie, Marburg
  - Klinikum der LMU München; Klinik und Poliklinik für Dermatologie und Allergologie, München
  - Klinikum rechts der Isar der TU München; Klinik & Poliklinik für Dermatologie und Allergologie, München
  - Universitätsklinikum Münster; Klinik für Hautkrankheiten; Allgemeine Dermatologie und Venerologie, Münster
  - Klinikum Nürnberg Nord; Hautklinik; Klinik für Dermatologie, Nuremberg
  - Harzklinikum Dorothea Christiane Erxleben GmbH; Klinik für Dermatologie und Allergologie, Quedlinburg
  - Universitätsklinikum Regensburg; Klinik und Poliklinik für Dermatologie, Regensburg
  - Universitaets-Hautklinik Tuebingen, Tübingen
  - Universitätsklinikum Würzburg; Klinik und Poliklinik für Dermatologie Venerologie u. Allergologie, Würzburg
- Greece (5):
  - Laiko General Hospital; 1St Pathological Clinic, Athens
  - Andreas Syggros Hospital; 1st University Dermatology Clinic; Oncology Department, Athens
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - University General Hospital of loannina; Dermatology and Venereal Diseases Clinic, Ioannina
  - Euromedical General Clinic of Thessaloniki; Oncology Department, Thessaloniki
- Hungary (5):
  - Semmelweis Egyetem; Bor-, Nemikortani es Boronkologiai Klinika, Budapest
  - Orszagos Onkologiai Intezet; B Belgyogyaszati Osztaly, Budapest
  - Debreceni Egyetem Klinikai Központ; Bőrgyógyászati Klinika, Debrecen
  - Kaposi Mor Teaching Hospital, Kaposvár
  - Szegedi Tud.Egyetem Szent-Gyorgyi Albert Klin.Kozp., Szeged
- Ireland (2):
  - Cork University Hospital; Dermatology Dept, Cork
  - St Vincent'S Uni Hospital; Medical Oncology, Dublin
- Israel (4):
  - Rambam Medical Center, Halfa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Sheba Medical Center; Tel Hashomer, Ramat Gan
- Italy (21):
  - Ospedale San Salvatore (ASL-01); Dip. di Dermatologia U.O.S. di Dermatologia Oncol, L’Aquila, Abruzzo
  - Ospedale Antonio Perrino; Oncologia Medica, Brindisi, Apulia
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Policlinico Sant'Orsola Malpighi; U.O. Dermatologia, Bologna, Emilia-Romagna
  - I.R.S.T. Srl - Meldola - FC; Day Hospital Oncologico, Meldola, Emilia-Romagna
  - Azienda Ospedaliera Umberto I; Clinica Dermatologica, Rome, Lazio
  - Fondazione Ptv Policlinico Tor Vergata; Dermatologia, Rome, Lazio
  - Istituto Dermatologico San Gallicano IRCCS; Dermatologia Oncolgica, Rome, Lazio
  - Istituto Dermopatico dell'Immacolata (IDI)-IRCCS; IV Divisione Oncologica e Dermatologia Oncologica, Rome, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Università di Brescia; Dipartimento di Dermatologia, Brescia, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori;S.S. Trattamento MedicoTumori dellaTesta e delCollo, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - IRCCS Istituto Clinico Humanitas; Farmacia, Rozzano, Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo; Dipartimento Oncologico, Candiolo, Piedmont
  - Ospedale Armando Businco; Dermatologia, Cagliari, Sardinia
  - A.O.U. Ospedali Riuniti Umberto I-G.M.Lancisi-G.Salesi Ancona;S.O.D. MED.Interna-Clinica Oncologica, Ancona, The Marches
  - Ospedale IOT- Palagi Dermatologia 2, Florence, Tuscany
  - A.O.U. Senese Policlinico Santa Maria Alle Scotte, Siena, Tuscany
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Seconda, Padua, Veneto
- National Cancer Institute, Vilnius, Lithuania
- Hospital General de México, Mexico City, Mexico CITY (federal District), Mexico
- Netherlands (4):
  - Academ Ziekenhuis Groningen; Medical Oncology, Groningen
  - LUMC; Dermatologie, Leiden
  - Maastricht University Medical Centre; Dermatologie, Maastricht
  - Erasmus MC; Dermatology, Rotterdam
- Waitemata District Health; General Surgery, Takapuna, New Zealand
- Oslo Universitetssykehus HF; Radiumhospitalet, Oslo, Norway
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - DERMED Centrum Medyczne; Sp zoo, Lodz
  - Centrum Diagnostyki Znamion, Poznan
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie; Klinika Onkologiczna, Warsaw
- IPO do Porto; Servico de Oncologia Medica, Porto, Portugal
- Romania (5):
  - Institutul Oncologic Prof. Dr. Al. Trestioreanu Bucuresti, Bucharest
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Oncology Center Sf. Nectarie, Craiova
  - Spital Clinic Judetean Mures; Oncologie, Târgu Mureş
  - S.C. Life Search S.R.L; Medical Oncology Clinic, Timișoara
- Russia (4):
  - FSBI"National Medical Research Center of Oncology named after N.N.Petrov" MHRF, Saint Petersburg, Sankt-Peterburg
  - FSBI "National Medical Research Center of Oncology N.N. Blokhin", Moscow
  - Moscow city oncology hospital #62 of Moscow Healthcare Department, Moscow
  - Saint-Petersburg City Clinical Oncology Dispensary, Saint Petersburg
- Serbia (2):
  - Institute for Oncology and Radiology of Serbia; Medical Oncology, Belgrade
  - Military Medical Academy, Belgrade
- Fakultna Nemocnica Roosevelta, Banská Bystrica, Slovakia
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- Spain (22):
  - Hospital Universitario Son Espases; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Hospital de Gran Canaria Dr. Negrin; Servicio de Dermatologia, Las Palmas de Gran Canaria, LAS Palmas
  - Fundacion Hospital de Alcorcon; Servicio de Dermatologia, Alcorcón, Madrid
  - Hospital Universitario del Sureste; Servicio de Dermatologia, Arganda, Madrid
  - Clinica Universitaria de Navarra; Servicio de Dermatologia, Pamplona, Navarre
  - Hospital Univ. Central de Asturias; Servicio de Dermatologia, Oviedo, Principality of Asturias
  - Complejo Hospitalario Nuestra Señora de la Candelaria; Servicio de Dermatologia, Santa Cruz de Tenerife, Tenerife
  - Hospital de Cruces; Servicio de Oncologia, Bilbao, Vizcaya
  - Hospital de la Santa Creu i Sant Pau; Servicio de Dermatologia, Barcelona
  - Hospital Clinic i Provincial; Servicio de dermatología, Barcelona
  - Hospital Reina Sofia; Servicio de dermatología, Córdoba
  - Hospital Universitario Virgen de las Nieves; Servicio de Oncologia, Granada
  - Hospital General Universitario de Guadalajara; Servicio de Dermatologia, Guadalajara
  - Complejo Asistencial Universitario de Leon; Servicio de Oncologia, León
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital General Universitario J.M Morales Meseguer; Servicio de Dermatologia, Murcia
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Complejo Hospitalario de Toledo- H. Virgen de la Salud; Servicio de Dermatologia, Toledo
  - Hospital General Universitario de Valencia; Servicio de oncologia, Valencia
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital Universitario Miguel Servet; Servicio Dermatologia, Zaragoza
- Sweden (2):
  - Skånes Onkologiska Klinik, Universitetssjukhuset, Lund
  - Karolinska Universitetssjukhuset, Solna, Stockholm
- Universitätsspital Zürich; Dermatologische Klinik, Zurich, Switzerland
- Turkey (Türkiye) (5):
  - Ankara Numune Training and Research Hospital; Dermatology, Ankara
  - Gazi Universitesi Tip Facultesi; Dept. of Dermatology, Ankara
  - Istanbul Uni of Medicine Faculty; Oncology Dept, Istanbul
  - Dokuz Eylul University Medicine Faculty; Dermatology, Izmir
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sıhhiye, Ankara
- United Kingdom (7):
  - Addenbrookes Hospital; Cambridge Cancer Trials Centre, S4 Box 279, Cambridge
  - Western Infirmary; Division of Cardiovascular and Medical Sciences, Glasgow
  - St Thomas Hospital, London
  - Royal Marsden Hospital - London, London
  - Freeman Hospital; Northern Centre For Cancer Care, New Castle Upon Tyne
  - Salford Royal NHS Foundation Trust, Salford
  - The Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Bossi P, Peris K, Calzavara-Pinton P, Queirolo P, Alfieri S, Palla M, Rossi MT, Spagnolo F, Tambone S, Astolfi C, Ascierto PA. Cohort analysis of safety and efficacy of vismodegib in Italian patients from the Phase II, multicenter STEVIE study. Future Oncol. 2020 Jun;16(16):1091-1100. doi: 10.2217/fon-2019-0664. Epub 2020 May 6. PMID 32374193
- [Derived] Basset-Seguin N, Hauschild A, Kunstfeld R, Grob J, Dreno B, Mortier L, Ascierto PA, Licitra L, Dutriaux C, Thomas L, Meyer N, Guillot B, Dummer R, Arenberger P, Fife K, Raimundo A, Dika E, Dimier N, Fittipaldo A, Xynos I, Hansson J. Vismodegib in patients with advanced basal cell carcinoma: Primary analysis of STEVIE, an international, open-label trial. Eur J Cancer. 2017 Nov;86:334-348. doi: 10.1016/j.ejca.2017.08.022. Epub 2017 Nov 5. PMID 29073584
- [Derived] Basset-Seguin N, Hauschild A, Grob JJ, Kunstfeld R, Dreno B, Mortier L, Ascierto PA, Licitra L, Dutriaux C, Thomas L, Jouary T, Meyer N, Guillot B, Dummer R, Fife K, Ernst DS, Williams S, Fittipaldo A, Xynos I, Hansson J. Vismodegib in patients with advanced basal cell carcinoma (STEVIE): a pre-planned interim analysis of an international, open-label trial. Lancet Oncol. 2015 Jun;16(6):729-36. doi: 10.1016/S1470-2045(15)70198-1. Epub 2015 May 13. PMID 25981813

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1232 participants were enrolled in the study, but only 1215 received at least one dose of any study treatment. Results include only the treated 1215 participants. Not Done category includes participants who did not complete the final end of study completion CRF page, including those who withdrew due to termination of the study.
Groups:
- Vismodegib - Locally Advanced; Vismodegib - Metastatic: Participants received vismodegib 150 mg orally once a day until one of the following occurred: Disease progression, intolerable toxicity most probably attributable to vismodegib, consent withdrawal, death, study termination by the Sponsor, or other reason deemed by the Investigator.
Period: Overall Study
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Started | 1119 | 96
Completed | 677 | 41
Not Completed | 442 | 55
Not completed — Death | 102 | 19
Not completed — Lost to Follow-up | 222 | 22
Not completed — Not Done | 118 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic | Total
Number analyzed (Participants) | 1119 | 96 | 1215
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (16.1) | 66.6 (13.0) | 69.5 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 485 | 36 | 521
  Male | 634 | 60 | 694
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Race data was not collected for participants enrolled from France as per local regulations.
  Participants
    Race: : Asian: number analyzed (Participants) | 1118 | 96 | 1214
    Race: : Asian | 1 | 0 | 1
    Race: : Black or African American: number analyzed (Participants) | 1118 | 96 | 1214
    Race: : Black or African American | 1 | 1 | 2
    Race: : White: number analyzed (Participants) | 1118 | 96 | 1214
    Race: : White | 787 | 92 | 879
    Race: : Other: number analyzed (Participants) | 1118 | 96 | 1214
    Race: : Other | 15 | 0 | 15
    Race: : Not Applicable: number analyzed (Participants) | 1118 | 96 | 1214
    Race: : Not Applicable | 314 | 3 | 317

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Any Adverse Events (AEs), AEs Grade 3 or 4, AEs Leading to Drug Interruptions or Discontinuations and Any Serious Adverse Events (SAEs)
Description: Adverse events were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activity of daily living with inability to perform bathing, dressing and undressing, feeding self, using the toilet, taking medications but not bedridden. Grade 4: An immediate threat to life. Urgent medical intervention is required in order to maintain survival.
Time Frame: Baseline to the data cut-off of 14 June 2017 (up to 6 years)
Measure: Number; unit: percentage of participants
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Number analyzed (Participants) | 1119 | 96
percentage of participants
  Any AEs | 98.4 | 99.0
  Any AEs with maximum severity of Grade 3 or 4 | 43.4 | 52.1
  Any Serious AEs | 24.3 | 32.3
  Any AEs leading to study drug interruption | 40.5 | 35.4
  Any AEs leading to study drug discontinuation | 33.8 | 17.7

2. Primary Outcome: Percentage of Participants Who Died Due to Adverse Events, Disease Progression or Other Reasons
Description: Reasons for "other" included "unknown," "natural causes," "cardiac decompensation," "general state alteration," "deterioration of general state," "clinical deterioration taking into consideration patient's age," "old age," and "disease progression of mediastinal squamous cell carcinoma (SCC)."
Time Frame: Baseline to the data cut-off of 14 June 2017 (up to 6 years)
Measure: Number; unit: percentage of participants
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Number analyzed (Participants) | 1119 | 96
percentage of participants
  Adverse Event | 6.1 | 6.3
  Disease Progression | 1.9 | 13.5
  Other | 1.3 | 0

3. Primary Outcome: Percentage of Participants Who Report a Shift in NCI CTCAE Grades to 3/4 in Hematology and Biochemistry Laboratory Parameters
Time Frame: Baseline to the data cut-off of 14 June 2017 (up to 6 years)
Measure: Number; unit: percentage of participants
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Number analyzed (Participants) | 1119 | 96
percentage of participants
  Hemoglobin (High) | 0.1 | 0
  Hemoglobin (Low) | 1.3 | 2.1
  Neutrophils, Total, Abs (Low) | 0.5 | 0
  Platelet (Low) | 0.2 | 0
  White Blood Cell Count (High) | 0.2 | 1.0
  White Blood Cell Count (Low) | 0.2 | 0
  Alkaline Phosphatase (High) | 0.6 | 0
  SGPT/ALT (alanine aminotransferase) - High | 2.2 | 4.2
  SGOT/AST (aspartate aminotransferase) - High | 1.5 | 3.1
  Creatine Kinase (High) | 0.1 | 0
  Creatinine (High) | 1.3 | 2.1
  Glucose (Low) | 0.4 | 0
  Potassium (High | 1.1 | 4.2
  Potassium (Low) | 0.8 | 1.0
  Sodium (High) | 0.2 | 0
  Sodium (Low) | 2.6 | 4.2
  Total Bilirubin (High) | 0.4 | 0

4. Primary Outcome: Exposure to Study Treatment: Duration on Treatment
Description: Duration on treatment was the number of days between first and last dose of study treatment.
Time Frame: Baseline to the data cut-off of 14 June 2017 (up to 6 years)
Measure: Median (Full Range); unit: days
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Number analyzed (Participants) | 1119 | 96
days | 256.0 [2 to 1904] | 337.0 [2 to 1932]

5. Primary Outcome: Exposure to Study Treatment - Dose Intensity
Description: Dose intensity was defined as the percentage of actual number of doses received versus planned.
Time Frame: Baseline to the data cut-off of 14 June 2017 (up to 6 years)
Measure: Median (Full Range); unit: percentage of doses
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Number analyzed (Participants) | 1119 | 96
percentage of doses | 97.62 [44.9 to 100.0] | 98.51 [67.8 to 100.0]

6. Secondary Outcome: Best Overall Response Rate (BORR)
Description: BORR was defined as the percentage of participants achieving either a complete response (CR) or a partial response (PR) as assessed by the Investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) required a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline to the data cut-off of 14 June 2017 (up to 6 years)
Population: Only included participants that had histologically confirmed measurable disease at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Number analyzed (Participants) | 1076 | 83
percentage of participants
  CR | 33.9 | 4.8
  PR | 35.3 | 32.5

7. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time interval between the date of the earliest qualifying response (CR or PR) and the date of disease progression or death for any cause. Median duration of response was estimated using Kaplan-Meier estimates.
Time Frame: Baseline to the data cut-off of 14 June 2017 (up to 6 years)
Population: Only included participants that had histologically confirmed disease, measureable disease status at baseline (measureable or non-measureable) and reported a response of CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Number analyzed (Participants) | 1103 | 89
months | 18.89 [17.64 to 22.57] | 13.93 [9.23 to 18.50]

8. Secondary Outcome: Time to Response
Description: Time to response was defined as the interval between the date of first treatment and the date of first documentation of confirmed CR or PR (whichever occur first).
Time Frame: Baseline to the data cut-off of 14 June 2017 (up to 6 years)
Population: Only included participants that had histologically confirmed measurable disease at baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Number analyzed (Participants) | 1076 | 83
months | 3.65 [2.92 to 3.71] | NA [5.49 to NA] — Not Estimated as the values were not estimable due to insufficient number of events.

9. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time interval between the date of the first therapy and the date of progression or death for any causes, whichever occurs first. Disease progression was assessed by the investigator.
Time Frame: Baseline to the data cut-off of 14 June 2017 (up to 6 years)
Population: Only included participants that had histologically confirmed disease and measureable disease status at baseline (measureable or non-measureable).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Number analyzed (Participants) | 1103 | 89
months | 20.30 [19.38 to 21.82] | 12.85 [11.30 to 17.68]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first treatment to the date of death, regardless of the cause of death.
Time Frame: Baseline to the data cut-off of 14 June 2017 (up to 6 years)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Number analyzed (Participants) | 1103 | 89
months | NA [NA to NA] — Median OS and 95% CI were not estimable due to low proportion of events. | NA [NA to NA] — Median OS and 95% CI were not estimable due to low proportion of events.

11. Secondary Outcome: Change From Baseline Scores of Skindex-16 Questionnaire Domains of Emotion, Function and Symptom
Description: The Skindex-16 questionnaire includes three domains for the assessment of the effects of skin disease on participants' quality of life: symptoms, emotions and function. For each domain, responses from the questionnaire were transformed to a linear scale of 100 varying from 0 (never bothered, i.e., best) to 100 (always bothers, i.e., worst).
Time Frame: Baseline to the data cut-off date of 14 June 2017 (up to 6 years).
Population: Only included participants that had histologically confirmed disease at baseline. For each time point, Number Analyzed refers to patients with non-missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
Number analyzed (Participants) | 1111 | 89
units on a scale
  Emotion: C2D1 (Cycle 2 Day 1): number analyzed (Participants) | 604 | 39
  Emotion: C2D1 (Cycle 2 Day 1) | -18.02 (26.12) | -8.68 (23.50)
  Emotion: C7D1: number analyzed (Participants) | 380 | 25
  Emotion: C7D1 | -26.04 (30.80) | -13.14 (33.25)
  Emotion: End of Study: number analyzed (Participants) | 335 | 18
  Emotion: End of Study | -24.66 (33.13) | 7.76 (27.61)
  Function: C2D1: number analyzed (Participants) | 603 | 39
  Function: C2D1 | -7.43 (22.18) | -1.71 (16.31)
  Function: C7D1: number analyzed (Participants) | 380 | 25
  Function: C7D1 | -11.09 (26.49) | -10.00 (24.74)
  Function: End of Study: number analyzed (Participants) | 334 | 18
  Function: End of Study | -9.84 (28.03) | 4.81 (29.80)
  Symptom: C2D1: number analyzed (Participants) | 604 | 39
  Symptom: C2D1 | -9.92 (22.02) | -5.06 (23.10)
  Symptom: C7D1: number analyzed (Participants) | 379 | 26
  Symptom: C7D1 | -12.03 (24.95) | -6.73 (28.92)
  Symptom: End of Study: number analyzed (Participants) | 334 | 18
  Symptom: End of Study | -11.85 (27.05) | 1.85 (22.15)

12. Secondary Outcome: Percentage of Participants With a ≥ 30% Reduction in Disease-Related Symptoms According to MDASI Scale
Description: M.D. Anderson Symptom Inventory (MDASI) scale. The MDASI core instrument is a 19-item patient self-report questionnaire whose items comprise two scales, symptom severity and symptom interference. For 13 items (i.e., pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, difficulty remembering things, lack of appetite, drowsiness, dry mouth, sadness, vomiting, and numbness or tingling), participants were asked to rate how severe the symptoms were when "at their worst" in the last 24 hours. For the remaining 6 items, participants were asked to rate how much the symptoms have interfered with 6 areas of functioning (i.e., general activity, walking, work, mood, relations with other people, and enjoyment of life) in the last 24 hours.
Time Frame: 08-May-2013 (Protocol Version ≥ 4) to the data cut-off date of 14 June 2017 (approximately 4 years and 1 month).
Population: Included only participants who were enrolled after Protocol Version 4 was implemented, had non-missing data and baseline score ≥4. Per protocol, the MDASI measurements were measured in Metastatic patients only.
Measure: Number; unit: Percentage of participants
Arm/Group | Vismodegib - Metastatic
Number analyzed (Participants) | 10
Percentage of participants | 60.0

13. Secondary Outcome: Percentage of Participants With a ≥ 30% Reduction in Composite Symptom Severity Score According to MDASI Scale
Description: as for outcome 12
Time Frame: 08-May-2013 (Protocol Version ≥ 4) to the data cut-off date of 14 June 2017 (approximately 4 years and 1 month).
Population: Included only participants who were enrolled after Protocol Version 4 was implemented, had non-missing data and average baseline score ≥ 4. Per protocol, the MDASI measurements were measured in Metastatic patients only.
Measure: Number; unit: Percentage of participants
Arm/Group | Vismodegib - Metastatic
Number analyzed (Participants) | 3
Percentage of participants | 33.3

ADVERSE EVENTS:
Time Frame: Baseline to the data cut-off of 14 June 2017 (up to 6 years)
Arm/Group | Vismodegib - Locally Advanced | Vismodegib - Metastatic
All-Cause Mortality (participants affected / at risk) | 103/1119 | 19/96
Serious Adverse Events (participants affected / at risk) | 272/1119 | 31/96
Other Adverse Events (participants affected / at risk) | 1065/1119 | 90/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib - Locally Advanced (N=1119) | Vismodegib - Metastatic (N=96)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 0
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0
LEFT VENTRICULAR DILATION (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 8 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 0
SINUS NODE DYSFUNCTION (Cardiac disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 3 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 3 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 0
VOLVULUS (Gastrointestinal disorders) | 0 | 1
PHARYNGO-OESOPHAGEAL DIVERTICULUM (Gastrointestinal disorders) | 1 | 0
ASTHENIA (General disorders) | 4 | 0
CHEST PAIN (General disorders) | 2 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 11 | 1
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 | 0
SUDDEN DEATH (General disorders) | 2 | 1
TERMINAL STATE (General disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 1
CHOLESTASIS (Hepatobiliary disorders) | 1 | 0
HEPATITIS (Hepatobiliary disorders) | 1 | 0
HEPATOTOXICITY (Hepatobiliary disorders) | 2 | 0
ABSCESS (Infections and infestations) | 2 | 0
APPENDICITIS (Infections and infestations) | 1 | 0
BACTERIAL INFECTION (Infections and infestations) | 1 | 0
BRAIN ABSCESS (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 2 | 0
CLOSTRIDIUM COLITIS (Infections and infestations) | 1 | 1
CYSTITIS (Infections and infestations) | 2 | 0
DIVERTICULITIS (Infections and infestations) | 2 | 0
ENDOCARDITIS BACTERIAL (Infections and infestations) | 1 | 0
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 5 | 1
GASTROENTERITIS CLOSTRIDIAL (Infections and infestations) | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1
GROIN ABSCESS (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 3 | 0
INFECTED SKIN ULCER (Infections and infestations) | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0
PNEUMONIA (Infections and infestations) | 17 | 1
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 3 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 1 | 0
EYEBALL AVULSION (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 8 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
FOREIGN BODY (Injury, poisoning and procedural complications) | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 6 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL INTESTINAL PERFORATION (Injury, poisoning and procedural complications) | 1 | 0
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 | 0
HEPATIC ENZYME INCREASED (Investigations) | 5 | 0
TRANSAMINASES INCREASED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 1 | 0
CACHEXIA (Metabolism and nutrition disorders) | 2 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 4 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 | 0
MUSCULOSKELETAL DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1
BREAST CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
LIP SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NON-SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 3 | 0
DIZZINESS (Nervous system disorders) | 1 | 1
DYSGEUSIA (Nervous system disorders) | 1 | 0
EMBOLIC STROKE (Nervous system disorders) | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 2 | 1
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 6 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
DISORIENTATION (Psychiatric disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 2 | 2
URETHRAL STENOSIS (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 4 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
ARTERIAL HAEMORRHAGE (Vascular disorders) | 1 | 0
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 0
HYPOTENSION (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0
BRONCHITIS (Infections and infestations) | 5 | 0
NORMOCHROMATIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
THROMBOCYTOMPENIA (Blood and lymphatic system disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 3 | 0
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 2 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 2 | 0
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 | 0
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0
PANCREATITIS (Gastrointestinal disorders) | 2 | 0
VOMITING (Gastrointestinal disorders) | 2 | 0
ABDOMINAL INCARCERATED HERNIA (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRIC PERFORATION (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 3 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
ILEUS (Gastrointestinal disorders) | 1 | 0
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0
ILL-DEFINED DISORDER (General disorders) | 2 | 0
PYREXIA (General disorders) | 2 | 0
CYST (General disorders) | 1 | 0
DEATH (General disorders) | 1 | 0
GAIT DISTURBANCE (General disorders) | 1 | 0
HERNIA (General disorders) | 1 | 0
IMPAIRED HEALING (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PAIN (General disorders) | 0 | 1
PERFORMANCE STATUS DECREASED (General disorders) | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 4 | 0
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 1 | 0
BILIARY COLIC (Hepatobiliary disorders) | 1 | 0
BILIARY CYST (Hepatobiliary disorders) | 1 | 0
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 | 0
HEPATIC MASS (Hepatobiliary disorders) | 1 | 0
HEPATITIS TOXIC (Hepatobiliary disorders) | 1 | 0
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 4 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 3 | 0
URINARY TRACT INFECTION (Infections and infestations) | 3 | 0
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 | 1
LUNG INFECTION (Infections and infestations) | 2 | 0
UROSEPSIS (Infections and infestations) | 2 | 0
ABSCESS LIMB (Infections and infestations) | 1 | 0
ACTINOMYCOSIS (Infections and infestations) | 1 | 0
ACUTE SINUSITIS (Infections and infestations) | 1 | 0
ENDOPHTHALMITIS (Infections and infestations) | 1 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0
GANGRENE (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 1 | 0
MENINGITIS BACTERIAL (Infections and infestations) | 1 | 0
MORGANELLA INFECTION (Infections and infestations) | 1 | 0
ORBITAL INFECTION (Infections and infestations) | 1 | 0
PERIORBITAL CELLULITIS (Infections and infestations) | 1 | 0
PNEUMONIA BACTERIAL (Infections and infestations) | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 | 0
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 0
BONE CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 1 | 0
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
CHEST INJURY (Injury, poisoning and procedural complications) | 1 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 1 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
WOUND SECRETION (Injury, poisoning and procedural complications) | 0 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 0
BLOOD TEST ABNORMAL (Investigations) | 1 | 0
EJECTION FRACTION DECREASED (Investigations) | 0 | 1
LIVER FUNCTION TEST INCREASED (Investigations) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 3 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
SOFT TISSUE MASS (Musculoskeletal and connective tissue disorders) | 1 | 0
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
MALIGNANT NEOPLASM OF EYELID (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BENIGN NEOPLASM OF ADRENAL GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
INVASIVE LOBULAR BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MARGINAL ZONE LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NASAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PAPILLARY RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RECTAL CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SKIN NEOPLASM BLEEDING (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 2 | 0
BRAIN OEDEMA (Nervous system disorders) | 1 | 0
CEREBROSPINAL FISTULA (Nervous system disorders) | 1 | 0
CEREBROVASCULAR DISORDER (Nervous system disorders) | 1 | 0
DEMENTIA (Nervous system disorders) | 1 | 0
FACIAL PARALYSIS (Nervous system disorders) | 0 | 1
FACIAL PARESIS (Nervous system disorders) | 1 | 0
FOCAL DYSCOGNITIVE SEIZURES (Nervous system disorders) | 1 | 0
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 1 | 0
LETHARGY (Nervous system disorders) | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 1
PARTIAL SEIZURES (Nervous system disorders) | 1 | 0
PRESYNCOPE (Nervous system disorders) | 1 | 0
SEIZURE (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0
TRIGEMINAL NEURALGIA (Nervous system disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 1
SOMATIC SYMPTOM DISORDER (Psychiatric disorders) | 1 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 3 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 | 0
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1 | 0
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SINUS POLYP (Respiratory, thoracic and mediastinal disorders) | 1 | 0
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
DERMAL CYST (Skin and subcutaneous tissue disorders) | 1 | 0
LICHEN SCLEROSUS (Skin and subcutaneous tissue disorders) | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 | 1
AORTIC ANEURYSM (Vascular disorders) | 0 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0
HAEMORRHAGE (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 | 0
THROMBOSIS (Vascular disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 2 | 0
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 1 | 0
DIPLOPIA (Eye disorders) | 1 | 0
LAGOPHTHALMOS (Eye disorders) | 1 | 0
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 | 0
DEVICE DISLOCATION (Product Issues) | 2 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0
EYELID OPERATION (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib - Locally Advanced (N=1119) | Vismodegib - Metastatic (N=96)
ABDOMINAL PAIN (Gastrointestinal disorders) | 78 | 8
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 64 | 6
CONSTIPATION (Gastrointestinal disorders) | 107 | 14
DIARRHOEA (Gastrointestinal disorders) | 183 | 18
NAUSEA (Gastrointestinal disorders) | 197 | 24
VOMITING (Gastrointestinal disorders) | 96 | 6
ASTHENIA (General disorders) | 276 | 19
FATIGUE (General disorders) | 185 | 16
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 55 | 6
WEIGHT DECREASED (Investigations) | 471 | 38
DECREASED APPETITE (Metabolism and nutrition disorders) | 283 | 23
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 117 | 9
BACK PAIN (Musculoskeletal and connective tissue disorders) | 53 | 7
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 754 | 62
AGEUSIA (Nervous system disorders) | 201 | 12
DIZZINESS (Nervous system disorders) | 66 | 9
DYSGEUSIA (Nervous system disorders) | 620 | 47
HEADACHE (Nervous system disorders) | 87 | 9
ALOPECIA (Skin and subcutaneous tissue disorders) | 700 | 50
PRURITUS (Skin and subcutaneous tissue disorders) | 61 | 9
OEDEMA PERIPHERAL (General disorders) | 34 | 5
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 54 | 6
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 52 | 7
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 59 | 10
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 55 | 5
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 31 | 8
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 49 | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 64 | 12
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 26 | 12
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 46 | 5
HYPERTENSION (Vascular disorders) | 58 | 6
MYALGIA (Musculoskeletal and connective tissue disorders) | 78 | 7
BLOOD CREATININE INCREASED (Investigations) | 31 | 6
ANAEMIA (Blood and lymphatic system disorders) | 81 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT01367665/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT01367665/SAP_001.pdf